CLINICAL TRIAL: NCT05111652
Title: Electromyographic Assessment of the Shoulder Stabilizing Musculature in CrossFit® Athletes. An Observational Analytical Study of Case-controls Prevalence
Brief Title: Electromyographic Assessment of the Shoulder Stabilizing Musculature in CrossFit® Athletes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Principal investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: CE012110
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Muscle Strain; Electromyography; Trapezius Muscle Strain
Keywords: Serratus muscle strain
MeSH Terms: conditions — Sprains and Strains | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — observational electromiographic musculature activation

SUMMARY:
This is an observational analytical study of prevalent cases and controls.

DETAILED DESCRIPTION:
Approximately 39 subjects who practice CrossFit at least 6 hours a week are invitated to participate in this observational study. It will measure the activation of trapezius and Serratus muscles by Electromyography experiencing a feeling of fatigue 7-8 in PushPress and PullUps.

ELIGIBILITY:
Inclusion Criteria:

* Practicing CrossFit® for at least 1 year
* A minimum of 6 hours per week CrossFit® training
* No shoulder pain at the time of measurement

Exclusion Criteria:

* Tendinitis
* Bursitis
* Sistematic disease
* Nurological disease
* Central or periferic disease

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes and amateurs who practice CrossFit® discipline, who have mastered the basic exercises of Pull-up and Push-Press.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Observation of Basal Activation in Trapezius and Serratus muscles and after Push-Press and Pull-Up exercises assessed by Electromyographic mDurance® | 10 minutes
  Trapezius and Serratus muscle activation analysis in CrossFit athletes with Electromyography system for the muscle activity assessment with the electrode tools

IPD SHARING:
Plan to Share IPD: No